CLINICAL TRIAL: NCT00003935
Title: Treatment of Children With Diffuse Intrinsic Brain Stem Glioma With Standard Dose Irradiation and Vincristine Plus Oral VP-16, A POG Pilot Study
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Children With Newly Diagnosed Brain Stem Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9836; POG-9836 (Other: Pediatric Oncology Group); CDR0000067127 (Other: Clinical Trials.gov); COG-P9836 (Other: Children's Oncology Group)
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Brain Tumors; Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms | interventions — Etoposide; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Induction: Patients receive oral etoposide daily on days 1-21 and vincristine sulfate IV on days 1, 8, and 15. Treatment repeats every 4 weeks for 2 courses. Patients receive radiation therapy daily for 6 weeks concurrently with induction chemotherapy. Maintenance: One week after induction therapy, patients receive vincristine sulfate IV on days 1 and 8 and oral etoposide daily on days 1-21. Treatment repeats every 4 weeks for 10 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter
  Interventions: Drug: etoposide; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: etoposide
  Other Names: VP-16; VePesid; NSC # 141540
Drug: vincristine sulfate
  Other Names: VCR; Oncovin; NSC # 067574
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vincristine plus etoposide and radiation therapy in treating children who have newly diagnosed brain stem glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of vincristine plus etoposide with concurrent radiotherapy on one year survival in children with newly diagnosed diffuse intrinsic brain stem glioma. II. Assess the toxicity of this regimen in this patient population.

OUTLINE: Induction: Patients receive oral etoposide daily on days 1-21 and vincristine IV on days 1, 8, and 15. Treatment repeats every 4 weeks for 2 courses. Patients receive radiotherapy daily for 6 weeks concurrently with induction chemotherapy. Maintenance: One week after induction therapy, patients receive vincristine IV on days 1 and 8 and oral etoposide daily on days 1-21. Treatment repeats every 4 weeks for 10 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed diffuse intrinsic brain stem glioma by MRI At least 2/3 of the tumor in the pons Tumor origin clearly in the pons At least 2 clinical features with less than 6 months duration: Cranial nerve deficit Long tract signs Ataxia No diffuse brain stem enlargement secondary to neurofibromatosis No diffuse leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 3 to 21 Performance status: Karnofsky or Lansky 50-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL ALT no greater than 5 times upper limit of normal Renal: Creatinine or GFR normal for age

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No other concurrent chemotherapy No prior chemotherapy Endocrine therapy: Prior glucocorticoids allowed Radiotherapy: No prior radiotherapy Surgery: No prior surgery Other: No other concurrent investigational drugs

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 1999-09; Primary Completion 2003-10 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year

SECONDARY OUTCOMES:
Monitor the toxicity

CONTACTS AND LOCATIONS:
Overall Officials: David N. Korones, MD, Study Chair — James P. Wilmot Cancer Center
Locations (110):
- United States (97):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Children's Hospital and Health Center, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Portland, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. John's Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - James H. Quillen College of Medicine, Johnson City, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Oncology P.A., Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - MBCCOP - South Texas Pediatric, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Roanoke Community Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Medical School-Charleston, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Royal Children's Hospital, Parkville, Victoria, Australia
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Clinique de Pediatrie, Geneva

REFERENCES:
- [Result] Korones DN, Fisher PG, Kretschmar C, Zhou T, Chen Z, Kepner J, Freeman C. Treatment of children with diffuse intrinsic brain stem glioma with radiotherapy, vincristine and oral VP-16: a Children's Oncology Group phase II study. Pediatr Blood Cancer. 2008 Feb;50(2):227-30. doi: 10.1002/pbc.21154. PMID 17278121